CLINICAL TRIAL: NCT03899870
Title: Factors Predicting Recurrence After Curative Resection for Rectal Cancer: a 16-year Study
Brief Title: Factors Predicting Recurrence in Rectal Cancer After Surgery
Status: Completed | Type: Observational
Sponsor: ammar houssem (Other)
Responsible Party: Sponsor-Investigator, ammar houssem, Surgeon, Université de Sousse
Organization: Université de Sousse (Other)
Other Study IDs: 654285
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Rectal Cancer; Rectal Adenocarcinoma
Keywords: rectal adenocarcinoma; recurrence; prognosis
MeSH Terms: conditions — Rectal Neoplasms; Recurrence | interventions — Proctectomy; Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Rectal resection — Patients underwent anterior or low anterior resection. Patients with tumors in the lower third of the rectum where anal sphincters could not be preserved underwent abdominoperineal resection. In majority of the cases, inferior mesenteric artery (IMA) was ligated caudal to the origin of the left colic artery. For the tumors of the upper rectum, partial excision of the mesorectum was performed up to the minimum of 5 cm from the inferior aspect of the tumor. For the tumors of the middle and low rectum a total mesorectum excision was done with the minimum distal mucosal margin of 1 to 2 cm. Ileostomy was performed in cases where colon was poorly prepared, anastomotic leak test was positive or colonel anastomosis was made. In most of the cases, open surgery was performed. Laparoscopic surgery was performed in selected cases. Wide local excision was performed in selected cases with T1 tumors without locoregional lymphadenopathy.
Drug: Neoadjuvant therapy — Patients with locally advanced disease (T3, T4) or lymph nodal positive disease were offered neoadjuvant therapy. In the neoadjuvant therapy, we used 45 Gy in 25 fractions with concurrent 5-fluorouracil [5-FU] and patients were operated 8 to 10 weeks after neoadjuvant therapy. In some cases, especially the elderly patients with multiple co-morbidities, we used short-course pelvic radiation therapy which included 25 Gy in 5 fractions over 1 week.
Drug: Adjuvant therapy — Patients with locally advanced disease (T3, T4) or lymph nodal positive disease were offered adjuvant therapy. In most of the cases, FOLFOX (leucovorin, 5-FU, oxaliplatin) regimen was used and for elderly patients who could not tolerated this regimen, we used oral capecitabine.

SUMMARY:
Colorectal cancer is one of the most frequently diagnosed cancers and a major cause of cancer deaths worldwide. Recurrence after curative surgery is one of the major factors affecting the long-term survival and its frequency is estimated to be 22.5% at 5 years. of which 12% have local recurrence. The overall survival in case of recurrence of 11% at 5 years.

Several patient-, tumor-related and treatment-related prognostic factors have been found to be associated with the risk of recurrence of rectal adenocarcinoma. Some of these factors such as TNM stage, lymphatic and perineural invasion and vascular emboli have been found to affect recurrence free survival in most studies. While the impact of other factors such as distal resection margin, tumor size, extra capsular spread and neoadjuvant chemoradiotherapy on recurrence remains controversial. Moreover, most of the previous studies on prognostic factors have been from American and European countries with very little data from African countries. Recognition of these factors helps in identification of high-risk patients who require close and more rigorous postoperative surveillance. Hence this study was conducted to determine the factors affecting recurrence after curative resection of rectal cancer in African population.

ELIGIBILITY:
Inclusion Criteria:

- all the patients who underwent curative resection for rectal adenocarcinoma between January 2000 and December 2015 at the Department of Digestive and Visceral Surgery of Sahloul Hospital, Sousse, Tunisia

Exclusion Criteria:

* patients who underwent palliative surgery
* patients with microscopically or macroscopically positive resection margin
* patients with tumors other than adenocarcinoma
* patients who died in the postoperative period due to complications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rectal adenocarcinoma who underwent curative resection
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Recurrence | through study completion at average of 5 years
  the development of any new malignant lesion within the field of surgery (locoregional recurrence) or outside it (distant metastasis) after initial resection was judged to be curative (R0) based on the preoperative imaging and histopathological examination of the resected specimen.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farhat W, Azzaza M, Mizouni A, Ammar H, Ben Ltaifa M, Lagha S, Kahloul M, Gupta R, Mabrouk MB, Ali AB. Factors predicting recurrence after curative resection for rectal cancer: a 16-year study. World J Surg Oncol. 2019 Oct 28;17(1):173. doi: 10.1186/s12957-019-1718-1. PMID 31660992